CLINICAL TRIAL: NCT01912391
Title: A Phase III Randomized Double-blind, 12 Week, Placebo Controlled Trial of Transdermal Selegiline in Borderline Personality Disorder (BPD) to Evaluate Efficacy and Safety
Brief Title: Clinical Research Study to Evaluate Selegiline in the Treatment of Borderline Personality Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mood and Anxiety Research, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PJM-01; WV26504-4245 (Other Grant/Funding Number: WV26504-4245)
Record Dates: First submitted 2013-07-16; First posted 2013-07-31 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Borderline Personality Disorder
Keywords: Depression; Anxiety; Headaches; Migraines; Irritable Bowel Syndrome IBS; Neurodermatitis; Fibromyalgia; Premenstrual Syndrome PMS; Temporomandibular Joint Dysfunction TMJ
MeSH Terms: conditions — Borderline Personality Disorder; Depression; Anxiety Disorders; Headache; Migraine Disorders; Irritable Bowel Syndrome; Neurodermatitis; Fibromyalgia; Premenstrual Syndrome | interventions — Selegiline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selegiline (Experimental): Transdermal Selegiline 12 mg patch Apply (1) patch daily
  Interventions: Drug: Selegiline
- Placebo (for Selegiline) (Placebo Comparator): Transdermal Placebo patch Apply (1) patch daily
  Interventions: Drug: Placebo (for Selegiline)

INTERVENTIONS:
Drug: Selegiline — The Study Drug known as either selegiline 12 mg patch or matching placebo patch will be administered daily beginning at Visit 2 for the duration of 12 weeks.
  Other Names: Emsam
  Arms: Selegiline
Drug: Placebo (for Selegiline) — Transdermal Placebo patch manufactured to mimic Transdermal Selegiline 12 mg. patch
  Arms: Placebo (for Selegiline)

SUMMARY:
Selegiline is superior to placebo in improving psychological and physical functioning in patients with Borderline Personality Disorder.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a chronic disorder occurring in 2-3% of the population. BPD is accompanied by high levels of co-existing psychiatric and physical disorders. One key predictor is persistent and recurring major depressive disorder.

Since BPD is most closely linked with mood disorders and depression in particular, the use of antidepressant medications to treat the disorder is logical. However, to date, there are no FDA approved treatments for BPD. The American Psychiatric Association's Treatment Guidelines for Borderline Personality Disorder recommend antidepressants as a primary treatment of the disorder.

Earlier trials using antidepressants that increase certain brain chemicals, such as, serotonin and noradrenalin have shown efficacy in controlling the mood swings of the illness for many people. These studies also document efficacy in controlling physical disorders, including headaches, migraines, irritable bowel, neurodermatitis (skin rash), fibromyalgia, premenstrual syndrome, and tempomandibular joint dysfunction (TMJ).

group of antidepressants known as monoamine oxidase inhibitors (MAOIs) have also been shown to be effective in BPD patients. The oral form of these medications was accompanied by dietary restrictions, potential drug interactions, blood pressure changes and weight gain.

Selegiline, a MAOI antidepressant, was put into a skin patch delivery system (transdermal) that reduced the side-effect profile. Trials without placebo control showed many individuals with BPD benefit from the selegiline skin patch. This trial will look at individuals on the selegiline and placebo to make sure the selegiline is or is not effective in treating BPD.

ELIGIBILITY:
Inclusion Criteria:

* Subject has primary diagnosis of Borderline Personality Disorder(BPD).
* Subject has Symptomatology of BPD for at least 1 year.
* Subject understands the study procedures and voluntarily agree to participate.
* Subject is able to read, understand and complete questionnaires.
* Subject agrees to use (2)acceptable forms of contraception throughout the study.
* Patient must have a screening SCL 90-R score of > 120 (range 0-360).

Exclusion Criteria:

* Subject is not pregnant or breast feeding.
* Subject is unlikely to adhere to the study procedures and restrictions.
* Patient has failed treatment due to lack of efficacy of monoamine oxidase inhibitor(MAOI) medication.
* Patient anticipates need for surgery during the study.
* Patient has another predominant personality disorder other than BPD.
* Subject has an active history of substance abuse or dependence, e.g.,Positive Drug screen
* Subject has other health issues which could interfere with study interpretation.
* Subject reports recent suicide attempts or homicide attempts in the past 3 months.
* Subject must be substance abuse or dependence clean for (1) year.
* Subject has a history of a primary malignancy < 5 yrs.
* Subject has a medical condition(s)that are excluded, per Protocol, or are unstable.
* Subject has abnormal screening laboratory values, per Protocol, or other clinically significant, unexplained laboratory abnormality.
* Subject is currently participating or has participated in a study within 30 days.
* Patient has donated blood products or has had phlebotomy of > 300 ml within 8 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Measurement: Changes in the Hopkins Symptom Checklist 90-Revised (SCL 90-R) scale | Weeks 1-12
  The study subject will complete the SCL 90-R questionnaire at each visit on arrival at the office prior to meeting with the research staff. This will serve as the primary efficacy measure of outcome for the study. This instrument has been utilized in clinical trials since the early 1960s, and has a good ability to measure overall levels of psychological and physical functioning in this patient group.

SECONDARY OUTCOMES:
Secondary Efficacy Measurement: Change in Hamilton Depression Inventory 17 Questions (HAM-D) | Weeks 1 - 12
  Clinician will administer the HAM-D scale to subject at each visit to assess any changes in their overall symptoms, functioning social and daily life.
Clinical Global Impression of Change- Clinician (CGIc) | Weeks 3-12
  Clinician will assess any improvement in their overall symptoms, functioning social and daily life beginning at week 3(Visit 3)through week 12 (Visit 6).
Clinical Global Impression Change- Patient (CGIp) | Weeks 3 -12
  Patient will assess any improvement in their overall symptoms, functioning social and daily life beginning at week 3(Visit 3)through week 12 (Visit 6).
Sheehan Disability Scale (SDS) | Weeks 1, 4, 12
  Patient will assess any improvement in their overall functioning in their work / school, social and daily life at 3 time points

OTHER OUTCOMES:
Clinical and Laboratory Measurements for Safety: Change in Columbia Suicide Severity Rating Scale (CSSRS); Adverse Events; Vitals Signs; Body Weight; Laboratory Values; Blood Pressure; Study Drug Compliance; Concomitant Medication Compliance | Treatment Phase (1-12 weeks)
  Study subjects will be monitored for safety throughout the study beginning at the Screening Visit (V1). At each visit, subjects will have various clinical, laboratory and safety measurements conducted. Results will be assessed by the clinical team and will be monitored, at each visit, until the term of their participation. A 2 week, post-study, follow-up will be conducted by the study staff.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Markovitz, MD, PhD, Study Director — Mood and Anxiety Research, Inc
Locations (1):
- Mood and Anxiety Research, Inc, Fresno, California, United States

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174